CLINICAL TRIAL: NCT03217110
Title: Cerebellar Transcranial Magnetic Stimulation and Cognitive Control
Brief Title: Cerebellar Stimulation and Cognitive Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Krystal Parker, PhD (Other)
Responsible Party: Sponsor-Investigator, Krystal Parker, PhD, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 201610712
Record Dates: First submitted 2017-06-30; First posted 2017-07-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Schizophrenia; Autism Spectrum Disorder; Bipolar Disorder; Depression; Parkinson Disease
Keywords: Cerebellum
MeSH Terms: conditions — Schizophrenia; Autism Spectrum Disorder; Bipolar Disorder; Depression; Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- patient active rTMS (Experimental): Subjects will receive 5 days of 2x daily rTMS targeted over the cerebellum.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- patient sham rTMS (Sham Comparator): Subjects will receive 5 days of 2x daily sham stimulation of the cerebellum.
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation (rTMS)
- Control active rTMS (Active Comparator)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Control sham rTMS (Sham Comparator)
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Subjects with neuropsychiatric diagnoses and matched-controls will be receive theta frequency stimulation of the cerebellum. We will target the cerebellar vermis.
  Other Names: rTMS
  Arms: Control active rTMS; patient active rTMS
Device: Sham Repetitive Transcranial Magnetic Stimulation (rTMS) — Subjects with neuropsychiatric diagnoses and matched-controls will be receive sham stimulation of the cerebellum. We will target the cerebellar vermis.
  Other Names: Sham stimulation
  Arms: Control sham rTMS; patient sham rTMS

SUMMARY:
The purpose of this study is to examine whether cerebellar stimulation can be used to improve cognitive deficits and mood in patients with schizophrenia, autism, bipolar disorder, Parkinson's disease, and major depression.

DETAILED DESCRIPTION:
Our recent work found that patients with Parkinson's disease and schizophrenia have impaired frontal EEG rhythms in the theta and delta range (1-8 Hz).We have been using transcranial direct current stimulation to recover these rhythms as patients perform elementary cognitive tasks. We found that although we are able to modulate cerebellar and frontal activity with tDCS, this effect is minimal as the depth of the current is not great enough to modulate all cerebellar activity. Here we use transcranial magnetic stimulation (TMS) to modulate neural activity in the frontal cortex and recover cognitive function in patients with autism, schizophrenia, bipolar disorder and Parkinson's disease.

The purpose of the study is to explore cerebellar stimulation as a potential new treatment to restore frontal activity and cognitive function in autism, schizophrenia, bipolar disorder and Parkinson's disease.Subjects will be brought in for 5 to 6 separate visits, with cerebellar or sham TMS stimulation twice per day for 5 days, as well as 3 follow-up visits.During these visits the patient will have cognitive, disease-specific and emotional testing, including EEG testing and MRI imaging. For those participants that received sham stimulation we will again use EEG to record how single pulses of magnetic or electrical stimulation influences other regions of the cerebellum and downstream brain regions. These data will provide insight into how the cerebellum may influence downstream brain regions and play a role in cognitive and motor performance. All data will be analyzed offline to determine if performance on the interval timing task and/or frontal brain rhythms change following transcranial magnetic stimulation as compared to the pre-stimulation blocks of trials. Additionally, we will analyze changes in their cognitive function, symptom ratings, functional and structural MRI, and mood following stimulation. Controls will receive both active and sham treatment for comparison.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis consistent with enrollment

Exclusion Criteria:

* History of recurrent seizures or epilepsy
* Any other neurological or psychiatric diagnosis outside the diagnosis for which the participant is enrolled.
* Active substance use disorder in the past 6 months other than tobacco use disorder.
* Inability to consent for study.
* Pacemaker
* Coronary Stent
* Defibrillator
* Neurostimulation
* Claustrophobia
* Uncontrolled high blood pressure
* Atrial fibrillation
* Significant heart disease
* Hemodynamic instability
* Kidney disease
* Pregnant, trying to become pregnant, or breast feeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-11-30 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in disease-specific symptom rating scale, one scale identified for each group (MADRS for bipolar group; PANSS for schizophrenia group; UPDRS in Parkinson's patient group). | During the 1 week of treatment, with follow up 1 week, 3 weeks, and 2 months post-stimulation.
  Change between pre- and post-assessments.

SECONDARY OUTCOMES:
Change in brain rhythms | During the 1 week of treatment, with follow up 1 week, 3 weeks, and 2 months post-stimulation.
  Change from baseline EEG activity in participants receiving stimulation during a timing task.
Change in cognitive function | During the 1 week of treatment, with follow up 1 week, 3 weeks, and 2 months post-stimulation.
  Improvement in cognitive function following cerebellar stimulation as compared to controls as measure by higher scores on an NIH Toolbox cognitive battery.
Changes in functional MRI | During the 1 week of treatment comparing pre- and post-stimulation scans.
  Changes in resting-state functional connectivity.
Change in NIH Toolbox emotion battery | During the 1 week of treatment, with follow up 1 week, 3 weeks, and 2 months post-stimulation.
  Improvement in emotion T-scores following cerebellar stimulation as compared to controls
Change in motor function | During the 1 week of treatment, with follow up 1 week, 3 weeks, and 2 months post-stimulation.
  Improvement in motor function as measured by the Abnormal Involuntary Movement Scale for schizophrenia patients.
Schizophrenia group: Change in Calgary depression scale. | During the 1 week of treatment, with follow up 1 week, 3 weeks, and 2 months post-stimulation.
  Improvement in Calgary depression scale from pre- to post-treatment assessments.
Bipolar group: Change in Young Mania Rating Scale. | During the 1 week of treatment, with follow up 1 week, 3 weeks, and 2 months post-stimulation.
  Improvement in YMRS scale from pre- to post-treatment.
Bipolar group: Change in Columbia Suicide Severity Rating Scale. | During the 1 week of treatment, with follow up 1 week, 3 weeks, and 2 months post-stimulation.
  Improvement in C-SSRS from pre- to post-treatment.
Change in PHQ9 score. | During the 1 week of treatment, with follow up 1 week, 3 weeks, and 2 months post-stimulation.
  Improvement in PHQ9 score from pre- to post-treatment.
Change in CGI. | During the 1 week of treatment, with follow up 1 week, 3 weeks, and 2 months post-stimulation.
  Improvement as measured on CGI from pre- to post-treatment.
Change in cognitive function. | During the 1 week of treatment, with follow up 1 week, 3 weeks, and 2 months post-stimulation.
  Improvements as measured by a neuropsychological battery pre and post-treatment.
Changes in structural MRI. | During the 1 week of treatment comparing pre- and post-stimulation scans.
  Changes in volumetrics in the active treatment group as compared to sham.
Changes in MRI-based timing task. | During the 1 week of treatment comparing pre- and post-stimulation scans.
  More accurate evaluation of a passage of time in the MRI scanner in the active treatment group as compared to the control group.
Changes in DTI. | During the 1 week of treatment comparing pre- and post-stimulation scans.
  Greater changes in the white matter tracts of the active treatment group as compared to the control group.
Changes in T1 rho MRI signal. | During the 1 week of treatment comparing pre- and post-stimulation scans.
  Normalization of T1 rho abnormalities greater in the active treatment group compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Krystal L Parker, Ph.D, Principal Investigator — Univeristy of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No